CLINICAL TRIAL: NCT06335082
Title: A Registry Based Collaborative to Measure Efficiency, Effectiveness, and Safety of Farapulse Pulsed Field Ablation Technology for Atrial Fibrillation
Brief Title: A Registry Based Collaborative to Measure Efficiency, Effectiveness, and Safety of Farapulse PFA Technology for AF
Acronym: DISRUPT-AF
Status: Enrolling by invitation | Type: Observational
Sponsor: Heart Rhythm Clinical and Research Solutions, LLC (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: DISRUPT-AF
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Atrial Fibrillation
Keywords: paroxysmal atrial fibrillation; persistent atrial fibrillation; long-standing persistent atrial fibrillation; pulse field ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- Acute Arm: Data will be collected at pre-ablation/baseline and at time of the ablation procedure. Sites should follow the subjects per their standard of care and at a minimum report any acute onset procedure or device-related complications through 30-days post procedure. Data collection will include procedural workflow, procedural outcomes, and acute onset procedure or device-related complications through 30 days.
  Interventions: Device: Pulsed Field Ablation
- Symptomatic Monitoring Only Arm (SMO): Data will be collected at pre-ablation/baseline, the ablation procedure, a 3-Month post-ablation office visit and 12-Months post-ablation (monitoring is triggered for symptomatic recurrences only). Data collection will include procedural workflow, procedural outcomes, acute, mid, and late onset procedure or device related complications, and symptomatic recurrence.
  Interventions: Device: Pulsed Field Ablation
- Full Monitoring Arm (FM): Data will be collected at pre-ablation/baseline, the ablation procedure, a 3-Month post-ablation office visit, interim continuous monitoring for asymptomatic arrhythmia recurrence at 6- and 12-Months post-ablation as well as monitoring as needed for symptomatic recurrences, and a 12-Month post-ablation office visit. Data collection will include procedural workflow, procedural outcomes, acute, mid, and late onset procedure or device related complications, symptomatic recurrence as well as asymptomatic recurrence.
  Interventions: Device: Pulsed Field Ablation

INTERVENTIONS:
Device: Pulsed Field Ablation — Ablation using the Boston Scientific Farapulse Pulsed Field Ablation System for the treatment of atrial fibrillation (AF)

SUMMARY:
The DISRUPT-AF Registry is an observational, prospective, multi-center, non-randomized, real-world registry designed to obtain clinical experience with the Farapulse Pulsed Field Ablation System for the treatment of atrial fibrillation (AF).

DETAILED DESCRIPTION:
The DISRUPT-AF Registry is an observational, prospective, multi-center, non-randomized, real-world registry designed to obtain clinical experience with the Farapulse Pulsed Field Ablation System for the treatment of atrial fibrillation (AF). All types of AF including paroxysmal, persistent and long standing persistent may be included.

The registry has three cohorts: 1) Acute Arm, 2) Symptomatic Monitoring Only Arm, and 3) Full Monitoring Arm. In the Acute Arm, patient assessments will occur at pre- procedure and procedure visits. In both the Symptomatic Monitoring Only Arm and the Full Monitoring Arm, patient assessments will occur at pre- procedure, procedure, 3 months, and 1 year post ablation. Additionally, the Full Monitoring Arm will assess for asymptomatic recurrence at 6- and 12-months post-ablation.

Sites will be assigned to an arm in which they will enroll under based on their practices current Standard of Care. Sites can only participate in one arm.

The primary purpose of the registry is to assess clinical outcomes, including procedural efficiency, safety, and long-term effectiveness of pulsed field ablation (PFA) in the treatment of patients with AF. Also, to assess the effect of PFA technology implementation on practice patterns, operational workflow and operator experience.

The registry will utilize real world clinical data obtained from the use of commercially available technologies under the authority of a health care practitioner within a legitimate practitioner-patient relationship.

ELIGIBILITY:
Inclusion Criteria:

* Patients who, in the opinion of the Investigator, are candidates for ablation for AF
* Plans to undergo an ablation procedure using the Farapulse Pulsed Field Ablation System manufactured by Boston Scientific
* De Novo ablation unless it is a repeat procedure for a subject whose index procedure is also included in the registry
* 18 years of age or older
* Able and willing to participate in baseline and follow up evaluations for the full length of the registry

Exclusion Criteria:

* Enrolled in an investigational drug or device trial, or any trial that dictates the treatment plan without prior approval from Sponsor
* Prior left atrial ablation (catheter or surgical)
* Currently receiving inotropic or mechanical support for Stage IV congestive heart failure, cardiogenic and/or septic shock.
* In the opinion of the Investigator, any known contraindication to an ablation procedure or to any device or drug required for use during an ablation procedure as assessed by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting at participating sites for atrial fibrillation ablation that meet all inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Long term effectiveness | 12 months
  Freedom from atrial arrhythmia recurrence post 90-day blanking period
Long-term safety | 12 months
  Rate of long-term safety events defined as procedure or device related reportable events (complications) that occur greater than 30 days post ablation. Data for this endpoint will be evaluated from the pooled results of the SMO and FM study arms.

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Arrhythmia Institute at Grandview, Birmingham, Alabama
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Community Memorial Health Systems, Ventura, California
  - The Arrythmia Center of South Florida, Delray Beach, Florida
  - Ascension St. Vincent's, Jacksonville, Florida
  - HCA Florida Mercy Hospital, Miami, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Endeavor Health (Northshore), Glenview, Illinois
  - Ascension St Vincent -Indianapolis Ascension Healt, Indianapolis, Indiana
  - MercyOne Iowa Heart Center, West Des Moines, Iowa
  - Norton Heart & Vascular Institute, Louisville, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Cardiovascular Associates of Delaware Valley, Haddon Heights, New Jersey
  - HCA Research Institute Mission Hospital, Asheville, North Carolina
  - The Christ Hospital - Heart & Vascular, Cincinnati, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - WellSpan Health, York, Pennsylvania
  - HCA - Trident Medical Center, North Charleston, South Carolina
  - Ascension St. Thomas Nashville, Nashville, Tennessee
  - Ascension Texas Cardiovascular, Austin, Texas
  - Texas Cardiac Arrhythmia Research Foundation (St. Davids), Austin, Texas
  - St. Mark's Hospital, Salt Lake City, Utah
  - HCA Research Institute - Chippenham Hospital, Richmond, Virginia

REFERENCES:
- [Derived] Al-Ahmad A, Osorio J, Day J, Wasserlauf J, Nair D, Eckart R, Campbell D, Dukes J, Cuoco F, Costello J, Zagrodzky J, Kessler D, Morales G, Rajendra A, Oza S, Barakat A, Magnano A, Amin A, Silverstein J, Thosani A, Bezenek SM, Zei P, Dai C, Natale A, Horton R; DISRUPT AF Investigators. Patient and Procedural Factors Associated With Same-Day Discharge Following Pulsed Field Ablation for Atrial Fibrillation: Insights From the DISRUPT-AF Registry. J Cardiovasc Electrophysiol. 2026 Jan;37(1):149-156. doi: 10.1111/jce.70210. Epub 2025 Dec 2. PMID 41331670